CLINICAL TRIAL: NCT04645784
Title: Investigating the Long-term Effect of Online Mental Health Literacy Training in Intercollegiate Sport
Brief Title: Long-term Effect of Online Mental Health Literacy Training
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Less participants than required
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, Laura Tennant, Principle Student Investigator, Brock University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: REB 20-091
Record Dates: First submitted 2020-11-18; First posted 2020-11-27 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Mental Health Literacy; Waitlist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Receives the supporting student-athlete mental wellness module
  Interventions: Other: Supporting Student-Athletes Mental Wellness
- Waitlist (No Intervention): Receives no intervention

INTERVENTIONS:
Other: Supporting Student-Athletes Mental Wellness — The module addresses: 1) managing your own mental wellness; 2) signs and symptoms of mental health problems; 3) role of student-athletes in creating a positive team environment that is supportive of mental health care seeking; 4) the role of a student-athlete in helping teammates; 5) how to identify emergency and non-emergency mental health situations.
  Arms: Intervention

SUMMARY:
The purpose of this study is to assess the effectiveness over time of an online mental health in sport module in improving mental health literacy, stigma, and help-seeking behaviors in a sample of Brock student-athletes. Student-athletes will be assigned to one of two conditions, mental health module or the waitlist condition. The mental health module will consist of completing the Supporting Student-Athletes Mental Wellness" online module for the student-athlete by the National Collegiate Athletics Association (NCAA). Participants will complete surveys at pre-intervention, post-intervention, 3-months and 6-month time points.

ELIGIBILITY:
Inclusion Criteria:

* student-athletes

Exclusion Criteria:

* non student-athletes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Multicomponent Mental Health Literacy Measure | 72 hours pre-intervention, 72 hours post-intervention, 3-months post, 6-months post
  Multicomponent Mental Health Literacy Measure
Change in Self-Stigma | 72 hours pre-intervention, 72 hours post-intervention, 3-months post, 6-months post
  Self Stigma of Seeking Help Survey
Change in Help seeking intentions | 72 hours pre-intervention, 72 hours post-intervention, 3-months post, 6-months post
  General Help-Seeking Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Philip Sullivan, Principal Investigator — Brock University
Locations (1):
- Brock University, St. Catharines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No